CLINICAL TRIAL: NCT01323205
Title: First-in-Patient Study to Assess the Safety and Tolerability and to Explore the Potential Therapeutic Efficacy of a Novel Glutamate Modulator as Monotherapy and as Add-On Therapy in Patients With Schizophrenia
Brief Title: Investigation of the Safety, Tolerability and Potential Therapeutic Effects of JNJ-40411813 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018340; 40411813SCH2001 (Other: Janssen Research & Development, LLC); 2010-023369-23 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: JNJ-40411813
MeSH Terms: conditions — Schizophrenia | interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-40411813 (Part A) (Experimental): JNJ-40411813 starting dose from 50 to 150 mg according to tolerability dose range increased stepwise from 50 mg to 150 mg capsule by mouth orally. Capsule (s) taken twice daily with a meal for 12 weeks.
  Interventions: Drug: JNJ-40411813
- JNJ-40411813 (Part B) (Experimental): JNJ-40411813 starting dose from 50 to 150 mg according to tolerability dose range increased stepwise from 50 mg to 150 mg capsule by mouth orally. Capsule (s) taken twice daily with a meal for 10 weeks.
  Interventions: Drug: JNJ-40411813; Drug: Antipsychotic medication
- Placebo and JNJ-40411813 (Part B) (Experimental): Placebo capsule (s) orally twice daily with a meal for 4 weeks followed by JNJ-40411813 according to tolerability dose range increased from 50 mg to 150 mg twice daily with a meal to 6 weeks.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Antipsychotic medication

INTERVENTIONS:
Drug: JNJ-40411813 — JNJ-40411813 starting dose from 50 to 150 mg according to tolerability dose range increased stepwise from 50 mg to 150 mg capsule by mouth orally. Capsule (s) taken twice daily with a meal for 12 weeks.
  Arms: JNJ-40411813 (Part A)
Drug: JNJ-40411813 — JNJ-40411813 starting dose from 50 to 150 mg as an add-on therapy. Dose is increased step-wise from 50 mg to 150 mg. Capsule(s) taken by mouth twice daily with a meal for 10 weeks.
  Arms: JNJ-40411813 (Part B); Placebo and JNJ-40411813 (Part B)
Drug: Placebo — Placebo capsule (s) orally twice daily with a meal for 4 weeks.
  Arms: Placebo and JNJ-40411813 (Part B)
Drug: Antipsychotic medication — Regular antipsychotic medications (Risperidone, Olanzapine, Clozapine, Amisulpride, Quetiapine, Paliperidone, Aripiprazole, Haloperidol, Levomepromazine, Zuclopenthixol Hydrochloride, Clotiapine, Pipamperone Hydrochloride, Benperidol, Flupentixol, Fluphenazine Decanoate, Melperone Hydrochloride, or Chlorpromazine Hydrochloride) will be continued in Part B.
  Arms: JNJ-40411813 (Part B); Placebo and JNJ-40411813 (Part B)

SUMMARY:
The purpose of this study is to explore the safety, tolerability, and potential clinical efficacy of JNJ 40411813 in schizophrenic patients.

DETAILED DESCRIPTION:
This is a first-in-human study of JNJ-40411813 in schizophrenic patients who are not currently receiving antipsychotic drug treatment (referred to as "(sub) acute" patients) and in patients who are currently taking antipsychotic drug treatment (referred to as "stable" patients). The study will consist of 2 parts: Part A and Part B. Part A will be open-label (patients will know the identity of study treatment), and (sub)acute schizophrenic patients will receive monotherapy (treatment with one drug) with JNJ-40411813. Part B will be double-blind (patient and study staff will not know the identity of study treatment) and will randomize (assign by chance) patients with stable but symptomatic schizophrenia to receive treatment with JNJ-40411813 or a placebo (treatment identical in appearance to JNJ-40411813 but does not contain active drug) as add-on therapy to their currently prescribed antipsychotic medication. Parts A (JNJ-40411813 monotherapy) and B (JNJ-40411813 add-on therapy) will run simultaneously. Patients will take JNJ-40411813 and placebo capsules orally (by mouth) twice daily (bid) with a meal. Part A: Patients will take JNJ-40411813 50 mg (1 capsule) bid up to 150 mg (3 capsules) bid for up to 12 weeks. Part B: Patients will take JNJ-40411813 50 mg bid or placebo bid for 4 weeks. After 4 weeks, the dose of JNJ-40411813 may be increased up to 150 mg bid for 6 weeks, and patients assigned to placebo may take JNJ-40411813 50 mg bid to 150 mg bid for up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 35 kg/m2 inclusive
* Medically stable on the basis of physical examination, medical history, vital signs, 12-lead ECG and clinical laboratory tests
* In- or outpatients who have been diagnosed with schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) at least 1 year prior to screening.

Exclusion Criteria:

* A current DSM-IV axis I diagnosis other than schizophrenia
* Any medical condition that could potentially alter the absorption, metabolism, or excretion of the study medication, such as Crohn's disease, liver disease, or renal disease
* Relevant history of any significant and/or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular disorders), renal, hepatic, endocrine, or immunologic diseases
* PANSS score <50 or >120
* Other significant and/or unstable systemic illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Udvalg for Klinische Undersogelser (UKU) ratings for side effects reported by patients | Up to 12 weeks
The number of patients with abnormal results from clinical laboratory tests performed as a measure of safety and tolerability | Up to 12 weeks
The number of patients with abnormal results from electrocardiograms (ECGs) performed as a measure of safety and tolerability | Up to 12 weeks
The number of patients with abnormal results from physical examinations (including vital signs measurements) performed as a measure of safety and tolerability | Up to 12 weeks
Number of patients with adverse events reported as a measure of safety and tolerability | Up to 12 weeks

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) scores to explore potential therapeutic effect of study drug | Up to 12 weeks
Clinical Global Impression - Schizophrenia (CGI-SCH) ratings to explore potential therapeutic effect of study drug | Up to 12 weeks
Subjective Well-being under Neuroleptics Scale (SWN) scores to explore potential therapeutic effect of study drug | Up to 12 weeks
Plasma (blood) concentration of JNJ-40411813 | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- Austria (3):
  - Innsbruck
  - Salzburg
  - Vienna
- Belgium (4):
  - Dave
  - Duffel
  - Kortenberg
  - Lede
- Bulgaria (2):
  - Plovdiv
  - Radnevo
- Germany (5):
  - Berlin
  - Hamburg
  - Mainz
  - Mannheim
  - München
- Romania (4):
  - Arad
  - Brasov
  - Iași
  - Sibiu
- Spain (2):
  - Barcelona
  - Zamora